CLINICAL TRIAL: NCT06999330
Title: Parcel-guided Transcranial Magnetic Stimulation for Anxiety in Parkinson's Disease
Brief Title: TMS in Anxiety-Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A25-040
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Parkinsons Disease (PD); Anxiety
Keywords: transmagnetic stimulation; functional MRI guided theta burst stimulation; intermittent theta burst stimulation
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Allocation ratio = 2:1 active intervention to sham.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Theta burst stimulation (Experimental): Subjects will receive treatment with intermittent theta burst stimulation (iTBS) with the active coil. There will be a total of 27 sessions over a 3-week period with 3 sessions per day. All subjects will receive iTBS to the left 8Av region. Total participation will be 8-12 weeks.
  Interventions: Device: Theta burst stimulation active coil
- Sham device (Sham Comparator): Subjects will receive treatment with sham coil. There will be a total of 27 treatments over a 3-week period. Coil will be placed over the same region as the experimental group. Total participation will be 8-12 weeks.
  Interventions: Device: Sham coil

INTERVENTIONS:
Device: Theta burst stimulation active coil — MagVenture TMS Therapy active coil with theta burst stimulation. Resting motor threshold: 90%; Number of pulses per session: 1200 pulses; Inter-train interval: 8 seconds; Pulse frequency in burst: 50 Hertz; Session length: 10 min; Time between sessions: 50 minutes.
  Other Names: Transmagnetic stimulation; MagVenture
  Arms: Theta burst stimulation
Device: Sham coil — MagVenture TMS Therapy sham coil
  Arms: Sham device

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease after Alzheimer's dementia. Anxiety in PD is common, has major effects on quality of life and contributes to increased disability. The reported prevalence of anxiety in PD ranges widely and is estimated up to 40%. Treatment with oral medications is not always effective or tolerated. TMS has been shown to be effective and safe in anxiety and general anxiety disorder (GAD), but there is only limited data available for Transcranial Magnetic Stimulation (TMS) treatment of anxiety in PD. Area 8Av is a parcellation based on Human connectome project within the left prefrontal cortex and is associated with GAD. Given the area's associations with mood disorders, its functional connectivity with large-scale brain networks involved in PD, and its anatomical accessibility by TMS, this may be an important target for anxiety in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Idiopathic PD defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor or rigidity and without any other known or suspected cause of Parkinsonism (according to MDS clinical diagnostic criteria for Parkinson's disease (42) Postuma et al, Movement Disorders 2015), confirmed by a fellowship trained movements disorder specialist.
2. Subject has a diagnosis of anxiety based on PAS (Parkinson's anxiety scale) score of ≥ 14
3. Subject is Hoehn & Yahr stage less than or equal to 3
4. Subject has a MOCA score ≥ 18
5. Subject is ≥ 40 and ≤ 90 years of age
6. Female subjects are post-menopausal or have a negative pregnancy test
7. The subject must be proficient in speaking, reading and understanding English in order to comply with procedural testing
8. Subject has provided informed written consent prior to participation. In the event that subject is legally unable to provide informed written consent due to deterioration in cognitive abilities, fully informed written consent must be provided by a legally authorized representative.
9. Subject is on a stable dose (at least 1 month prior to baseline visit) of antiparkinsonian agents and is willing to remain on this dose for the duration of the study. If the subject is on a anti-depressant or anti-anxiety medication, a stable dose without changes for 1 month is also required.

Exclusion Criteria:

1. Inability to tolerate imaging; contraindication of imaging due to implants or metal. This includes an implanted deep brain stimulation device.
2. Seizure disorder, active alcohol or substance use disorder.
3. Inability to speak and read English.
4. Anything else that, in the opinion of the PI/Clinician, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
5. Subject has atypical Parkinson's syndrome(s) due to drugs (e.g., metoclopramide, neuroleptics), metabolic neurogenetic disorders (e.g., Wilson's Disease), encephalitis, cerebrovascular disease, or degenerative disease (e.g., Progressive Supranuclear Palsy, Multiple System Atrophy, Corticobasal Degeneration, Lewy Body dementia)
6. Other forms of advanced dementia (PDD, AD), or MOCA <18
7. Subject has history of any of the following: moderate to severe pulmonary disease, poorly controlled congestive heart failure, significant cardiovascular and/or cerebrovascular events within previous 6 months, or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator.
8. Subject has history of any psychiatric illness that would pose a safety risk to the subject as determined by investigator.
9. Subject is currently taking sedative medications that are clinically contraindicated as determined by investigator.
10. Subject has undergone a recent change (<1 month) in their anti-parkinsonian medication, or anti-depressant medication or anti-anxiety medication at the baseline visit.
11. Safety risk to the subject as determined by investigator.
12. Subject has participated in a clinical trial investigation within 3 months of this study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | screening
  Percentage of participant who enroll and consent based on those contacted. A higher percentage indicates higher feasibility.
Participation Rate | 3 weeks
  Percentage of participant who start treatment after enrollment. A higher percentage indicates higher feasibility.
Fidelity | 2 weeks
  Percentage of participant who complete all treatment sessions. A higher percentage indicates higher fidelity.
Completion Rate | 2 weeks
  Percentage of participant who complete 7 of the 9 treatment visits. A higher percentage indicates higher completion.
Adverse Events Rate - Safety | up to 12 weeks
  Percentage of participant with adverse events. A lower percentage indicates a safer treatment.
Adverse Events Safety | up to 12 weeks
  Frequency of each adverse event. A higher frequency indicates a less safe treatment.

SECONDARY OUTCOMES:
Average change between baseline and 1 week post-treatment TMS vs Sham - Anxiety Scale | baseline, 1 week post-treatment
  The Parkinson Anxiety Scale (PAS) is a 12-item scale developed to assess anxiety in individuals with Parkinson's disease (PD). Items are scored on a 5 point Likert scale. Range [0-48]. A higher score indicates higher anxiety
Average change between baseline and 1 week post-treatment TMS vs Sham - Cognitive scale | baseline, 1 week post-treatment
  The Montreal Cognitive Assessment (MoCA) is a brief cognitive screening measure that has been validated for use among individuals with Alzheimer's disease. The total score for this test is 30 points, but one point will be added for individuals with ≤ 12 years of education. The cutoff point for normal cognition is 26/30 in the general population and in individuals with Parkinson's Disease. This will be conducted by clinical staff and gathered as part of the chart review. Range: [0-30]. Higher score indicates higher cognitive health.
Average change between baseline and 1 week post-treatment TMS vs Sham - Mood | baseline, 1 week post-treatment
  The Geriatric depression scale (GDS-15) short form is a screening measure for depression in older patients. Range [0-15]. A higher score indicates more depressive symptoms.
Average change between baseline and 1 week post-treatment TMS vs Sham - Motor | baseline, 1 week post-treatment
  The United Parkinson's Disease Rating Scale (UPDRS) is the most widely used clinical rating scale for Parkinson's disease. Only part III of the rating scale is used, which is a clinician-scored monitored motor evaluation, allowing ratings from 0 (no symptoms) to 4 (severe symptoms) for each Parkinson's motor symptom. The Movement Disorders Society (MDS) commissioned a revision of the scale, resulting in a new version, termed the MDS sponsored UPDRS revision (MDS-UPDRS). In this study, the MDS-UDPRS version will be used. Range [7-86]. A higher score indicates more severe motor symptoms.
Pre-post change between baseline and 1 week post-treatment within individuals in active TMS group - Anxiety Scale | baseline, 1 week post-treatment
  The Parkinson Anxiety Scale (PAS) is a 12-item scale developed to assess anxiety in individuals with Parkinson's disease (PD). Items are scored on a 5 point Likert scale. Range [0-48]. A higher score indicates higher anxiety
Pre-post change between baseline and 1 week post-treatment within individuals in active TMS group - Cognitive scale | baseline, 1 week post-treatment
  The Montreal Cognitive Assessment (MoCA) is a brief cognitive screening measure that has been validated for use among individuals with Alzheimer's disease. The total score for this test is 30 points, but one point will be added for individuals with ≤ 12 years of education. The cutoff point for normal cognition is 26/30 in the general population and in individuals with Parkinson's Disease. This will be conducted by clinical staff and gathered as part of the chart review. Range: [0-30]. Higher score indicates higher cognitive health.
Pre-post change between baseline and 1 week post-treatment within individuals in active TMS group - Mood | baseline, 1 week post-treatment
  The Geriatric depression scale (GDS-15) short form is a screening measure for depression in older patients. Range [0-15]. A higher score indicates more depressive symptoms.
Pre-post change between baseline and 1 week post-treatment within individuals in active TMS group - Motor | baseline, 1 week post-treatment
  The United Parkinson's Disease Rating Scale (UPDRS) is the most widely used clinical rating scale for Parkinson's disease. Only part III of the rating scale is used, which is a clinician-scored monitored motor evaluation, allowing ratings from 0 (no symptoms) to 4 (severe symptoms) for each Parkinson's motor symptom. The Movement Disorders Society (MDS) commissioned a revision of the scale, resulting in a new version, termed the MDS sponsored UPDRS revision (MDS-UPDRS). In this study, the MDS-UDPRS version will be used. Range [7-86]. A higher score indicates more severe motor symptoms.
Responder Rate | baseline, 1 week post treatment
  Percentage of participants that respond to treatment based on improvement in symptom specific scales. Higher percentage indicates more successful treatment

OTHER OUTCOMES:
Explore the effect of TMS treatment on functional connectivity with Left 8 Av. - Change | baseline, 1-week post treatment
  Average change between baseline and 1-week post-treatment will be compared between groups (TMS vs Sham) in anomaly burden.
Explore the effect of TMS treatment on functional connectivity with Left 8 Av. - Names and number of anomalous parcellations | baseline, 1-week post treatment
  Names and number of anomalous parcellations identified using connectivity analysis at baseline and 1-week post treatment will be described for each participant and tabulated for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with other researchers.